CLINICAL TRIAL: NCT03006172
Title: A Phase I, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0077 as a Single Agent in Patients With Locally Advanced or Metastatic PIK3CA-Mutant Solid Tumors and in Combination With Endocrine and Targeted Therapies in Patients With Locally Advanced or Metastatic PIK3CA-Mutant Breast Cancer
Brief Title: To Evaluate the Safety, Tolerability, and Pharmacokinetics of Inavolisib Single Agent in Participants With Solid Tumors and in Combination With Endocrine and Targeted Therapies in Participants With Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO39374; 2016-003022-17 (EudraCT Number); 2023-508124-36-00 (Other: EU CT Number)
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Solid Tumor
Keywords: PIK3CA mutant, Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — inavolisib; Fulvestrant; Letrozole; palbociclib; Metformin; Trastuzumab; pertuzumab

ARMS (9):
- Stage I Arm A: Inavolisib Single Agent (Experimental): Participants will receive inavolisib in escalating dose levels with starting dose of 6 milligrams (mg). Participants will receive single dose of inavolisib on Day 1 of Cycle 1 followed by once daily from Day 8 of Cycle 1. (Cycle length: 35 days for Cycle 1 and 28 days for all other cycles). Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib
- Stage I Arm B: Inavolisib + Palbociclib + Letrozole (Experimental): Participants will receive inavolisib in escalating dose levels (starting dose 3 mg) on Days 1-28, palbociclib on Days 1-21, and letrozole on Days 1-28 of each 28-day cycle. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Letrozole; Drug: Palbociclib
- Stage I Arm C: Inavolisib + Letrozole (Experimental): Participants will receive inavolisib in escalating dose levels along with letrozole on Days 1-28 of each 28-day cycle. The starting dose of inavolisib will not exceed the starting dose in Stage I Arm A. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Letrozole
- Stage II Arm B: Inavolisib + Palbociclib + Letrozole (Experimental): Participants will receive inavolisib on Days 1-28 in combination with palbociclib on Days 1-21 and letrozole on Days 1-28 of each 28-day cycle. Dose of inavolisib will be decided based on the results of Stage I Arm B. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Letrozole; Drug: Palbociclib
- Stage II Arm C: Inavolisib + Letrozole (Experimental): Participants will receive inavolisib in combination with letrozole on Days 1-28 of each 28-day cycle. Dose of inavolisib will be decided based on the results of Stage I Arm C. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Letrozole
- Stage II Arm D: Inavolisib + Fulvestrant (Experimental): Participants will receive inavolisib on Days 1-28 in combination with fulvestrant on Day 1 and 15 of Cycle 1 and then on Day 1 from Cycle 2 (cycle length: 28 days). Dose of inavolisib will be decided based on the results of Stage I Arm C. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant
- Stage II Arm E: Inavolisib + Palbociclib + Fulvestrant (Experimental): Participants will receive inavolisib (Days 1-28) in combination with palbociclib (Days 1-21) and fulvestrant (Days 1 and 15 of Cycle 1; Day 1 for subsequent cycles)(Cycle = 28 days). Dose of inavolisib will be determined from the results of Stage I Arm B. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant; Drug: Palbociclib
- Stage II Arm F: Inavolisib + Palbociclib + Fulvestrant + Metformin (Experimental): Participants will receive inavolisib (Days 1-28) in combination with palbociclib (Days 1-21), fulvestrant (Days 1 and 15 of Cycle 1; Day 1 for subsequent cycles) and metformin (Days 1-28)(Cycle = 28 days). Dose of inavolisib will be determined from the results of Stage I Arm B. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Fulvestrant; Drug: Palbociclib; Drug: Metformin
- Stage II Arm G: Inavolisib + Trastuzumab + Pertuzumab (Experimental): Participants will receive inavolisib in combination with trastuzumab and pertuzumab (Days 1-21). Dose of inavolisib will be determined from the results of Stage I Arm A. Participants will continue treatment until the end of the study in the absence of unacceptable toxicities and unequivocal disease progression.
  Interventions: Drug: Inavolisib; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Inavolisib — Participants will receive oral inavolisib once daily on Days 1-28 of each 28-day cycle (Arms A, B, C, D, E, F) or Days 1-21 of each 21-day cycle (Arm G).
  Other Names: RO7113755, GDC-0077
Drug: Fulvestrant — Participants will receive fulvestrant 500 mg, administered intramuscularly on Days 1 and 15 of Cycle 1. For subsequent cycles, participants will receive fulvestrant intramuscularly on Day 1 of each cycle.
  Arms: Stage II Arm D: Inavolisib + Fulvestrant; Stage II Arm E: Inavolisib + Palbociclib + Fulvestrant; Stage II Arm F: Inavolisib + Palbociclib + Fulvestrant + Metformin
Drug: Letrozole — Participants will receive once daily oral doses of letrozole 2.5 mg on Days 1-28 of each cycle.
  Arms: Stage I Arm B: Inavolisib + Palbociclib + Letrozole; Stage I Arm C: Inavolisib + Letrozole; Stage II Arm B: Inavolisib + Palbociclib + Letrozole; Stage II Arm C: Inavolisib + Letrozole
Drug: Palbociclib — Participants will receive once daily oral doses of palbociclib 125 mg on Days 1-21 of each cycle.
  Arms: Stage I Arm B: Inavolisib + Palbociclib + Letrozole; Stage II Arm B: Inavolisib + Palbociclib + Letrozole; Stage II Arm E: Inavolisib + Palbociclib + Fulvestrant; Stage II Arm F: Inavolisib + Palbociclib + Fulvestrant + Metformin
Drug: Metformin — Participants will receive oral metformin once daily, starting on Cycle 1, Day 1, as tolerated.
  Arms: Stage II Arm F: Inavolisib + Palbociclib + Fulvestrant + Metformin
Drug: Trastuzumab — Participants will receive trastuzumab, administered by IV infusion on Day 1 of each 21-day cycle, at a loading dose of 8 mg/kg for Cycle 1 and a dose of 6 mg/kg for subsequent cycles, until disease progression or unacceptable toxicity.
  Arms: Stage II Arm G: Inavolisib + Trastuzumab + Pertuzumab
Drug: Pertuzumab — Participants will receive pertuzumab, administered by IV infusion on Day 1 of each 21-day cycle, at a loading dose of 840 mg for Cycle 1 and a dose of 420 mg for subsequent cycles, until disease progression or unacceptable toxicity.
  Arms: Stage II Arm G: Inavolisib + Trastuzumab + Pertuzumab

SUMMARY:
This is an open-label, multicenter, Phase I study designed to evaluate the safety, tolerability, and pharmacokinetics of inavolisib administered orally as a single agent in patients with locally advanced or metastatic PIK3CA-mutant solid tumors, including breast cancer, and in combination with standard-of-care endocrine and/or targeted therapies for the treatment of locally advanced or metastatic PIK3CA-mutant breast cancer. Participants will be enrolled in two stages: a dose-escalation stage (Stage I) and an expansion stage (Stage II). Participants will be assigned to one of seven regimens: inavolisib as a single agent (Arm A), inavolisib in combination with palbociclib and letrozole (Arm B), inavolisib in combination with letrozole (Arm C), inavolisib in combination with fulvestrant (Arm D), inavolisib in combination with palbociclib and fulvestrant (Arm E), inavolisib in combination with palbociclib, fulvestrant, and metformin (Arm F), and inavolisib in combination with trastuzumab and pertuzumab (and letrozole or fulvestrant, if applicable (Arm G)).

ELIGIBILITY:
Inclusion Criteria:

* Evaluable or measurable disease per RECIST, Version 1.1 (measurable disease only for Arm D)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy of greater than or equal to (>=) 12 weeks
* Adequate hematologic and organ function, including blood counts, liver and kidney function

Stage I Arm A (Inavolisib):

- Locally advanced, recurrent, or metastatic, PIK3CA mutant, incurable solid tumor malignancy, including breast cancer

Stages I and II, Arms B and C:

- Postmenopausal female participants with locally advanced or metastatic PIK3CA-mutant HR+/HER2- breast cancer

Stage II, Arms D, E, or F:

- Female participants with locally advanced or metastatic PIK3CA-mutant HR+/HER2- breast cancer

Stage II Arm D:

- Prior treatment with CDK4/6 inhibitor

Stage II Arm G:

* Female participants with locally advanced or metastatic PIK3CA-mutant HER2+ breast cancer
* Left ventricular ejection fraction 50% or greater

Stages I and II:

- All participants must provide tumor tissue from the primary or metastatic tumor site obtained from a prior or new biopsy or surgical procedure for detection of PIK3CA mutation by central laboratory test.

Exclusion Criteria:

* Metaplastic breast cancer
* History of leptomeningeal disease
* Type 1 or 2 diabetes requiring anti-hyperglycemic medication
* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known and untreated, or active central nervous system metastases
* Uncontrolled pleural effusion or ascites
* Any active infection that could impact patient safety or serious infection requiring intravenous antibiotics
* History of other malignancy within 5 years, except for treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* History of or active ventricular dysrhythmias or congestive heart failure requiring medication or symptomatic coronary heart disease
* Congenital long QT syndrome, prolonged QT interval, or family history of sudden unexplained death or long QT syndrome

Stage II Arms B, C, D, and E only:

* Prior treatment with >1 chemotherapy regimen for metastatic disease
* Prior treatment with PI3K inhibitor
* History of significant toxicity related to mTOR inhibitor requiring treatment discontinuation

Stage II Arms B and E only:

- Prior CDK4/6 inhibitor treatment

Stage II Arm G only:

* Current uncontrolled hypertension or unstable angina
* History of congestive heart failure, serious cardiac arrhythmia, or recent myocardial infarction
* Prior ejection fraction decrease on trastuzumab
* Prior cumulative doxorubicin greater than 360 mg/m2
* Symptomatic active lung disease
* History of significant toxicity related to trastuzumab and/or pertuzumab requiring discontinuation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Percentage of Participants With Dose Limiting Toxicities | Day 1 up to Day 28 (for Stage 1 Arm A: Day 1 up to Day 35)
Recommended Phase II Dose of Inavolisib | Day 1 up to Day 28 (for Stage 1 Arm A: Day 1 up to Day 35)
Percentage of Participants With Adverse Events and Serious Adverse Events | Day 1 up to 6 years

SECONDARY OUTCOMES:
Area Under the Concentration Time-Curve (AUC) from Time Zero to Infinity (AUCinf) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to end of study (EOS; up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
AUC from Time Zero to Dosing Interval (AUC0-tau) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Half-Life of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Maximum Plasma Concentration (Cmax) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Minimum Plasma Concentration (Cmin) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Time to Cmax (tmax) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Apparent Clearance (CL/F) of Inavolisib | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
Accumulation Ratio (AR) of Inavolisib at Steady-State | Predose (0-2 hours before dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days (Cycle 1 of Stage 1 Arm A=35 days)
AUC of Palbociclib | Predose (0-2 hours before inavolisib) dosing) on Cycle 1 Day 1 up to Cycle 6; Cycle length=28 days
Cmax of Palbociclib | Predose (0-2 hours before inavolisib) dosing) on Cycle 1 Day 1 up to Cycle 6; Cycle length=28 days
AUC of Letrozole | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days
Cmax of Letrozole | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days
AUC of Fulvestrant | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days
Cmax of Fulvestrant | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=28 days
Percentage of Participants With Objective Response as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 (v1.1) | Baseline up to occurrence of complete response (CR) or partial response (PR) on 2 consecutive occasions >/=4 weeks apart (up to approximately 6 years)
Duration of Response, as Assessed by RECIST v1.1 | From first occurrence of a documented objective response (CR or PR) to disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Percentage of Participants With Clinical Benefit as Assessed by RECIST v1.1 | Baseline up to disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Progression Free Survival (PFS) as Assessed by RECIST v1.1 | Baseline up to disease progression or death from any cause, whichever occurs first (up to approximately 6 years)
Change in Maximum Standard Uptake Value (SUV) of Tumor Regions of Interest (as assessed by [18] F-fluorodeoxyglucose-positron emission tomography) From Baseline to Approximately 2 Weeks of Inavolisib Treatment | Baseline, Week 2
AUC of Pertuzumab | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=21 days
Cmax of Pertuzumab | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=21 days
AUC of Trastuzumab | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=21 days
Cmax of Trastuzumab | Predose (0-2 hours before inavolisib dosing) on Cycle 1 Day 1 up to EOS (up to approximately 6 years); Cycle length=21 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- United States (4):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (2):
  - Institut Bergonie, Bordeaux
  - Institut Gustave Roussy, Villejuif
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- United Kingdom (3):
  - Royal Marsden Hospital - Surrey, Surrey, Sutton
  - St Bartholomew's Hospital, London
  - Royal Marsden Hospital - London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jhaveri KL, Accordino MK, Bedard PL, Cervantes A, Gambardella V, Hamilton E, Italiano A, Kalinsky K, Krop IE, Oliveira M, Schmid P, Saura C, Turner NC, Varga A, Cheeti S, Hilz S, Hutchinson KE, Jin Y, Royer-Joo S, Peters U, Shankar N, Schutzman JL, Juric D. Phase I/Ib Trial of Inavolisib Plus Palbociclib and Endocrine Therapy for PIK3CA-Mutated, Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced or Metastatic Breast Cancer. J Clin Oncol. 2024 Nov 20;42(33):3947-3956. doi: 10.1200/JCO.24.00110. Epub 2024 Sep 5. PMID 39236276